CLINICAL TRIAL: NCT04639297
Title: NeruoVision Versus Standard Hospital Neuromonitoring, Influence on the Rate of Neurologic Injury Following Spine Surgery? A Randomized Controlled Trial
Brief Title: NeuroVision vs Standard Neuromonitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kern Singh, MD, Professor, Attending Physician, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19121607
Record Dates: First submitted 2019-12-17; First posted 2020-11-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Neurologic Deficits
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NeuroVision® IONM (Experimental): Patients scheduled to undergo a primary single or multilevel lateral spinal surgery procedures for non-trauma condition. Use of NeuroVision® IONM in lateral spine surgery to provide real-time visible and auditory tcMEP and CMAP waveforms.
  Interventions: Device: NeuroVision® IONM
- Conventional hospital based IONM (Active Comparator): Patients scheduled to undergo a primary single or multilevel lateral spinal surgery procedures for non-trauma condition. Use of hospital based IONM in lateral spine surgery to provide real-time visible and auditory tcMEP and CMAP waveforms.
  Interventions: Device: Hospital Based IONM

INTERVENTIONS:
Device: NeuroVision® IONM — Using NeuroVision® prior to surgery SSEP and tcMEP and values are recorded. A deficit of SSEP tracking is defined as an amplitude reduction of more than 10% or a latency increase more than 50%. Similarly, a CMAP amplitude reduction demonstrates problematic tcMEP monitoring.
  Arms: NeuroVision® IONM
Device: Hospital Based IONM — Using hospital based IONM prior to surgery SSEP and tcMEP and values are recorded. A deficit of SSEP tracking is defined as an amplitude reduction of more than 10% or a latency increase more than 50%. Similarly, a CMAP amplitude reduction demonstrates problematic tcMEP monitoring.
  Arms: Conventional hospital based IONM

SUMMARY:
The purpose of this study is to perform a prospective, randomized, controlled clinical trial to assess the utility of IONM in patients undergoing primary, single or multilevel lateral spinal procedures. Subjects will be randomized to undergo a lateral spine surgery with the use of NeuroVision® IONM or conventional hospital based IONM to assess incidence of new-onset neurological injury.

DETAILED DESCRIPTION:
Elective spinal surgery for the correction of degenerative spinal pathology may involve significant intraoperative risks that can influence postoperative neurologic outcomes. Spinal cord monitoring had made it possible to track the spine and nerve root sensory and motor tracts. This has improved the ability to conduct minimally invasive surgery by allowing surgeons to operate without direct visualization of the neurologic elements.

Intraoperative neuromonitoring (IONM) of the spinal cord is primarily accomplished by both somatosensory evoked potentials (SSEP) and transcranial motor evoked potentials (tcMEPs). Due to a shortage in personnel trained to evaluate neuro-monitoring results, surgeon-driven systems have been established. An example of a surgeon driven monitoring system is NeuroVision®, which interacts with the surgeon during the operation by providing real-time visible and auditory tcMEP and compound muscle action potential (CMAP) waveforms. This stands in comparison to hospital based methods of IONM.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary single or multilevel lateral spinal surgery procedures for degenerative pathology Diagnosis: myelopathy, radiculopathy, myeloradiculopathy, central stenosis, foraminal stenosis herniated nucleus pulposus, degenerative disc disease, spondylosis, and osteophytic complexes
* Patients able to provide informed consent

Exclusion Criteria:

* Active infection
* Active or history of malignancy
* Spinal traumatic injury within the past 2 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of new-onset neurological injury | Enrollment up to 2 years postoperatively
  Decreased somatosensory evoked potentials (SSEP) and transcranial MEPs (tcMEPs)

SECONDARY OUTCOMES:
Cost analysis of IONM use | Enrollment up to 1 month post-operative
  Difference in costs of hospital IONM and Neurovision
False positive and false negative events in each modality | Intraoperatively up to 1 day post-operative
  Incorrect labeling of SSEP, tcMEP, and surface electromyography (sEMG) signals
Adverse Events | Postoperative to documented progress assessed up to 2 months
  Post-operative nausea and vomiting, Gastro-esophageal reflux, ileus, urinary tract infection, venous thromboembolic events, Respiratory depression/airway compromise,m renal insufficiency, wound complications

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No